CLINICAL TRIAL: NCT03176004
Title: Attention Training to Modify Error-related Negativity and Risk for Anxiety in Adolescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Greg Hajcak, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MH106477
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Adolescents are randomized to either a game that trains attention away from threat (attention bias modification), a game that trains attention but unrelated to threat (control condition), or a wait list group.
Who Masked: Participant, Investigator
Masking Description: Research assistants assign participants to condition; the investigator is unaware of the assignment. Participants are unaware of the distinction between ABM and CC, though they would know if they were in the wait list group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Bias Modification (Experimental): Participants play a game in which they can move up in levels by reducing their reaction time to targets presented in the location of a threatening word.
  Interventions: Other: Attention Bias Modification
- Active Control Condition (Active Comparator): Participants play a game in which they can move up in levels by reducing their reaction time to targets presented in the location of a word with a specific color.
  Interventions: Other: Attention Bias Modification
- Wait List (No Intervention): Participants simply return after 8 weeks.

INTERVENTIONS:
Other: Attention Bias Modification — A computer game is used to facilitate attention away from threatening words.
  Arms: Active Control Condition; Attention Bias Modification

SUMMARY:
This is a multi-site study to examine error-related brain activity (i.e., the error-related negativity) and anxiety symptoms in 11 to 14 year-olds (N=600) at two time points separated by two years. The study examines the degree to which error-related negativity can predict anxiety prospectively over two years, and whether a computerized game that alters attention to threat can alter error-related negativity and trajectories of anxiety.

DETAILED DESCRIPTION:
Approximately 600 youths between the ages of 11 and 14 and their parents will be assessed. Adolescents will be evaluated at baseline using event-related potentials, self-report, and interview-based measures. The error-related negativity will be evaluated immediately (it takes less than 5 minutes to process and score a single subjects' error-related negativity ), and adolescents with good error-related negativity data (~90%, based on scorable error-related negativity data) will be randomly assigned to either an 8-week (i.e., 16 session) adaptive attention bias modification (N=180) or control condition (N=180) or a waitlist condition (N=180) group. Each session lasts 20 minutes, and participants will be asked to complete two 20-minute sessions per week. Participants will be assessed immediately at post, using the same measures from the baseline assessment. All participants will complete a 2-year follow-up lab visit using the same measures from the baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

* children and parent must speak English well enough to complete the study assessments

Exclusion Criteria:

* current threat of harm to self or others, bipolar illness, psychosis, thought disorder, pervasive developmental disorder, mental retardation, neurological diseases that impair cognition, or significant head injuries (past 3 months).

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Symptoms | Baseline to 8 week
  Symptoms of Anxiety on the Screen for Child Anxiety Related Emotional Disorders (SCARED)
Change in Anxiety Symptoms | baseline to 2 year follow-up
  Symptoms of Anxiety on the Screen for Child Anxiety Related Emotional Disorders (SCARED)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - San Diego State University, San Diego, California
  - Florida State University, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: Yes
Data is being uploaded to the Research Domain Criteria Database, and will be available through National Institute of Mental Health Data Archive; the analyzed data yielded in our project, as specified in the same document (i.e., 12 months after accomplishment of each primary aim or objective, or immediately upon publication of the project's primary results, whichever occurs first).